CLINICAL TRIAL: NCT07342530
Title: Early Intervention for Postpartum PTSD: Comparing Written Exposure and Capnometry Guided Breathing Therapy
Brief Title: Early Support for Post-Traumatic Stress Disorder After Difficult Childbirth: Writing and Breathing Interventions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Arkansas (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Pervez Sultan, Professor of Anesthesiology, Perioperative and Pain Medicine (Obstetrics), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80498; R01AT013866-01 (NIH)
Record Dates: First submitted 2026-01-09; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Written Exposure Therapy; Breathing Techniques; PTSD (Childbirth-Related); Postpartum Care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Postpartum Standard of Care (No Intervention): Participants will follow their current standard of care.
- Written Exposure Therapy (WET) (Experimental): Participants will complete 5 writing sessions focused on their childbirth experience. One 50-minute session will be held in the hospital before discharge, followed by four 50-minute sessions by secure video once a week. Sessions are delivered by a trained study therapist under licensed clinician supervision.
  Interventions: Behavioral: Written Exposure Therapy (WET)
- Capnometry-Guided Breathing Intervention (CGRI) (Experimental): Participants will complete one 45-minute in-hospital training session using the device, which includes a tablet and breathing sensor. They will then practice guided breathing at home twice daily for about 17 minutes each time for 4 weeks, with weekly phone check-ins from study staff.
  Interventions: Device: Capnometry-Guided Breathing Intervention (CGRI)

INTERVENTIONS:
Behavioral: Written Exposure Therapy (WET) — Participants will complete 5 writing sessions focused on their childbirth experience. One 50-minute session will be held in the hospital before discharge, followed by four 50-minute sessions by secure video once a week. Sessions are delivered by a trained study therapist under licensed clinician supervision.
  Arms: Written Exposure Therapy (WET)
Device: Capnometry-Guided Breathing Intervention (CGRI) — Participants will complete one 45-minute in-hospital training session using the device, which includes a tablet and breathing sensor. They will then practice guided breathing at home twice daily for about 17 minutes each time for 4 weeks, with weekly phone check-ins from study staff.
  Other Names: Freespira
  Arms: Capnometry-Guided Breathing Intervention (CGRI)

SUMMARY:
The purpose of this study is to examine two early interventions, Written Exposure Therapy and Capnometry Guided Breathing, to reduce post-traumatic stress disorder (PTSD) symptoms in women after childbirth as compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Delivered a live infant within 5 days
* Severe maternal morbidity or infant admitted to NICU
* PCL-5 ≥28
* English-speaking
* Able to consent and participate

Exclusion Criteria:

* Active psychosis or mania
* Current suicidal crisis
* Current suicidal intent or plan
* Cognitive impairment preventing participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 70 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants initiating assigned treatment | Baseline (up to 2 weeks)
  Proportion of participants who begin their assigned intervention (≥1 session for WET; completion of initial training for CGRI)
Percentage of participants completing Written Exposure Therapy (WET) | Baseline to Week 6
Percentage adherence to Written Exposure Therapy (WET) | Baseline to Week 6
Percentage of participants completing Capnometry Guided Respiratory Intervention (CGRI) | Baseline to Week 6
Percentage adherence to Capnometry Guided Respiratory Intervention (CGRI) | Baseline to Week 6
Participant Satisfaction Scale Score using Client Satisfaction Questionnaire (CSQ-8) | Week 5
  Participant satisfaction measured using the CSQ-8 questionaire, an 8-item scale. (Scale score 8 - 32. Higher scores represent greater satisfaction with treatment.)
Treatment credibility using the Opinion About Treatment (OAT) form | Week 5
  Participant perceptions of treatment credibility will be measured using the OAT form. (Scale score 3 - 27. Higher scores represent greater perceived credibility of the intervention.)

SECONDARY OUTCOMES:
Change from baseline in PTSD Checklist for DSM-5 (PCL-5) Scale Score | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 12
  Change in PTSD symptoms during past week measured by the PTSD Checklist for DSM-5 (PCL-5), a 20-item self-report measure. (Score range 0 - 80, higher scores indicating greater severity of PTSD symptoms.).
Change from baseline in Edinburgh Postnatal Depression Scale (EPDS) Scale Score | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 12
  Participants complete the EPDS questionnaire, a 10-item scale assessing postpartum depressive symptoms over the past 7 days. (Score range 0 - 30, higher scores represents greater symptom severity.)
Change from baseline in Whole Person Health Index (WPHI) Scale Score | Baseline, Week 3, Week 6, Week 12
  Participants complete WHPI questionaire, a 9 item scale assessing global health and functioning. (Score range 9 - 81, higher scores represent better health).
Change from baseline in Generalized Anxiety Disorder Questionaire (GAD-7) | Baseline, Week 3, Week 6, Week 12
  Participants complete the GAD-7, a 7-item scale assessing anxiety symptoms over 2 weeks. (Score range 0 - 21, higher scores represent greater anxiety severity.)
Change from baseline in Maternal-infant bonding (MIBS) Scale Score | Baseline, Week 3, Week 6, Week 12
  Participants complete the MIBS questionaire, an 8 item measure of bonding difficulties over the past few weeks (Score range 0 - 24, higher scores represent greater bonding impairment).
Change from baseline in STanford Obstetric Recovery checKlist (STORK) scale score | Baseline, Week 3, Week 6, Week 12
  Participants complete the STORK questionnaire, a 47-item scale assessing postpartum recovery over the past 7 days. (Score range 0 - 188, higher score represents a greater degree of recovery)
Change from baseline in Breastfeeding Self-Efficacy Scale-Short Form (BFSES-SF) | Baseline, Week 3, Week 6, Week 12
  Participants complete the BFSES-SF, a 14-item measure of breastfeeding self-efficacy (Score range 14 - 70, higher scores indicate greater breastfeeding confidence.)
Percentage of participants completing hair sample collection at Baseline and Week 6 | Baseline, Week 6
  Participants have hair samples collected at baseline and at Week 6 post treatment.
Change in hair cortisol concentration between Baseline and Week 6 | Baseline, Week 6
  Participants have hair samples collected at baseline and at Week 6 post treatment. Hair steroid concentrations reflect average systemic hormone exposure over the preceding weeks. Change in hair cortisol concentration from Baseline to Week 6
Change in hair cortisone concentration between Baseline and Week 6 | Baseline, Week 6
  Participants have hair samples collected at baseline and at Week 6 post treatment. Hair steroid concentrations reflect average systemic hormone exposure over the preceding weeks. Change in hair cortisone concentration from Baseline to Week 6
Change in hair testosterone concentration between Baseline and Week 6 | Baseline, Week 6
  Participants have hair samples collected at baseline and at Week 6 post treatment. Hair steroid concentrations reflect average systemic hormone exposure over the preceding weeks. Change in hair testosterone concentration from Baseline to Week 6
Change in hair progesterone concentration between Baseline and Week 6 | Baseline, Week 6
  Participants have hair samples collected at baseline and at Week 6 post treatment. Hair steroid concentrations reflect average systemic hormone exposure over the preceding weeks. Change in hair progesterone concentration from Baseline to Week 6
Change in hair corticosterone concentration between Baseline and Week 6 | Baseline, Week 6
  Participants have hair samples collected at baseline and at Week 6 post treatment. Hair steroid concentrations reflect average systemic hormone exposure over the preceding weeks. Change in hair corticosterone concentration from Baseline to Week 6
Change in hair dehydroepiandrosterone (DHEA) concentration between Baseline and Week 6 | Baseline, Week 6
  Participants have hair samples collected at baseline and at Week 6 post treatment. Hair steroid concentrations reflect average systemic hormone exposure over the preceding weeks. Change in hair dehydroepiandrosterone (DHEA) concentration values from Baseline to Week 6
Change in hair androstenedione concentration between Baseline and Week 6 | Baseline, Week 6
  Participants have hair samples collected at baseline and at Week 6 post treatment. Hair steroid concentrations reflect average systemic hormone exposure over the preceding weeks. Change in hair androstenedione concentration from Baseline to Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Pervez Sultan, Principal Investigator — Stanford University; Debra Kaysen, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University, Palo Alto, California

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Wish whom? Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. For what types of analysis? For individual participant data meta-analysis By what mechanism will data be made available? Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be provided).